CLINICAL TRIAL: NCT03474081
Title: A Phase IV, 12 Week, Randomised, Double-blind, Double-dummy Study to Compare Single Inhaler Triple Therapy, Fluticasone Furoate/Umeclidinium/Vilanterol (FF/UMEC/VI), With Tiotropium Monotherapy Based on Lung Function and Symptoms in Participants With Chronic Obstructive Pulmonary Disease
Brief Title: A Comparative Study Between Fluticasone Furoate/Umeclidinium/Vilanterol (FF/UMEC/VI) Single Inhaler Triple Therapy Versus Tiotropium Monotherapy in Subjects With Chronic Obstructive Pulmonary Disease (COPD)
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Collaborators: Parexel (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 207626; 2017-001190-16 (EudraCT Number)
Record Dates: First submitted 2018-03-15; First posted 2018-03-22 (Actual); Results first posted 2020-04-24 (Actual); Last update posted 2021-07-15 (Actual); Status verified 2021-07

CONDITIONS: Pulmonary Disease, Chronic Obstructive
Keywords: Umeclidinium; Lung function; RESPIMAT; Chronic obstructive pulmonary disease; Triple Therapy; Vilanterol; HANDIHALER; Tiotropium; Fluticasone furoate
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — Tiotropium Bromide; Albuterol

STUDY DESIGN:
Intervention Model Description: Subjects will be randomized 1:1 to receive either FF/UMEC/VI via ELLIPTA DPI along with placebo to match tiotropium or tiotropium via HANDIHALER along with placebo to match FF/UMEC/VI in the morning for 84 days.
Who Masked: Participant, Investigator
Masking Description: This will be a double blind study. Subjects and investigator will be masked.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: Yes

ARMS (2):
- Subjects receiving FF/UMEC/VI + Placebo to match tiotropium (Experimental): Eligible subjects will receive FF/UMEC/VI at a dose of 100/62.5/25 microgram (mcg) administered once daily in the morning via ELLIPTA along with placebo to match tiotropium administered once daily in the morning via HANDIHALER. Subjects will self-administer 4 puffs of rescue medication (Albuterol/salbutamol) via metered dose inhaler (MDI).
  Interventions: Drug: FF/UMEC/VI; Drug: Albuterol/salbutamol; Drug: Placebo to match tiotropium; Device: ELLIPTA inhaler; Device: HANDIHALER; Device: MDI
- Subjects receiving Tiotropium + Placebo to match FF/UMEC/VI (Experimental): Eligible subjects will receive Tiotropium at a dose of 18 mcg administered once daily in the morning via HANDIHALER along with placebo to match FF/UMEC/VI administered once daily in the morning via ELLIPTA. Subjects will self-administer 4 puffs of rescue medication (Albuterol/salbutamol) via MDI.
  Interventions: Drug: Tiotropium; Drug: Albuterol/salbutamol; Drug: Placebo to match FF/UMEC/VI; Device: ELLIPTA inhaler; Device: HANDIHALER; Device: MDI

INTERVENTIONS:
Drug: FF/UMEC/VI — A single inhaler triple therapy of FF/UMEC/VI will be provided via ELLIPTA DPI. FF/UMEC/VI will be available as dry white powder with dosing strengths of 100/25/62.5 mcg per blister.
  Arms: Subjects receiving FF/UMEC/VI + Placebo to match tiotropium
Drug: Tiotropium — Tiotropium will be provided as a hard gelatin capsule for oral inhalation containing 18 mcg tiotropium bromide blended with lactose, administered via HANDIHALER DPI.
  Arms: Subjects receiving Tiotropium + Placebo to match FF/UMEC/VI
Drug: Albuterol/salbutamol — Albuterol/salbutamol will be provided as an inhalation via MDI with a spacer or nebules and will be given as a rescue medication throughout the study.
Drug: Placebo to match FF/UMEC/VI — Placebo matching FF/UMEC/VI will be available as a dry white powder of lactose or magnesium stearate, administered via ELLIPTA DPI.
  Arms: Subjects receiving Tiotropium + Placebo to match FF/UMEC/VI
Drug: Placebo to match tiotropium — Placebo will be given as hard gelatin capsule for oral inhalation containing lactose, administered via HANDIHALER DPI.
  Arms: Subjects receiving FF/UMEC/VI + Placebo to match tiotropium
Device: ELLIPTA inhaler — ELLIPTA DPI will contain two individual blister strips with 30 blisters per strip. FF/UMEC/VI and placebo to match FF/UMEC/VI will be administered to the subjects using ELLIPTA DPI.
Device: HANDIHALER — Tiotropium and placebo to match tiotropium will be administered to the subjects using HANDIHALER DPI.
Device: MDI — Albuterol/salbutamol will be provided as a rescue medication throughout the study using MDI.

SUMMARY:
COPD is a progressive disease characterized by increasing obstruction to airflow and the progressive development of respiratory symptoms including chronic cough, increased sputum production, dyspnea and wheezing. Once-daily triple therapy of an Inhaled Corticosteroid/ Long-acting Muscarinic Receptor Antagonists/ Long Acting Beta-Agonist (ICS/LAMA/LABA) that is combination of FF/UMEC/VI in a single device is being developed with the aim of providing a new treatment option for the management of advanced COPD. The primary purpose of this study is to evaluate lung function and health related quality of life (HRQoL) after 84 days of treatment with a single inhaler triple therapy combination of FF/ UMEC/VI once daily via the ELLIPTA® dry powder inhaler (DPI) compared with tiotropium once daily via HANDIHALER®, in subjects with COPD. Subjects will be randomized 1:1 to receive FF/UMEC/VI or tiotropium in the morning for 84 days. Subjects will also receive albuterol/salbutamol as a rescue therapy throughout the study. Approximately 848 subjects with advanced COPD will be enrolled in the study. The total study duration will be approximately 17 weeks including, 4-week run-in period, 12-week treatment period and a 1-week follow-up period. ELLIPTA is a registered trademark of GlaxoSmithKline (GSK) group of companies. HANDIHALER and RESPIMAT are registered trademarks of Boeringher Ingelheim.

ELIGIBILITY:
Inclusion Criteria:

* Subjects capable of giving signed informed consent.
* Outpatients will be included in the study.
* Subjects 40 years of age or older at Screening (Visit 1).
* Male or female subjects will be included; a female subject is eligible to participate if she is not pregnant, not breastfeeding, and at least one of the following conditions applies: not a woman of childbearing potential (WOCBP) or a WOCBP who agrees to follow the contraceptive guidance during the treatment period and until the safety follow-up contact after the last dose of study treatment.
* An established clinical history of COPD in accordance with the definition by the American Thoracic Society/European Respiratory Society.
* Current or former cigarette smokers with a history of cigarette smoking of >=10 pack-years at Screening (Visit 1) (number of pack years = [number of cigarettes per day / 20] x number of years smoked [example given {e.g.}, 20 cigarettes per day for 10 years, or 10 cigarettes per day for 20 years]). Previous smokers are defined as those who have stopped smoking for at least 6 months prior to Visit 1.
* A score of >=10 on the COPD Assessment Test (CAT) at Screening (Visit 1).
* Subjects must demonstrate at Screening: A post-bronchodilator FEV1 <50 percent predicted normal or a post-bronchodilator FEV1 <80 percent predicted normal and a documented history of >=2 moderate exacerbations or one severe (hospitalized) exacerbation in the previous 12 months. Subjects must also have a measured post albuterol/salbutamol FEV1/forced vital capacity (FVC) ratio of <0.70 at screening.
* Subjects must have been receiving daily maintenance treatment with tiotropium alone (via the HANDIHALER or RESPIMAT®) for their COPD for at least 3 months prior to Screening.

Exclusion Criteria:

* Women who are pregnant or lactating or are planning on becoming pregnant during the study.
* Subjects with a current diagnosis of asthma. (Subjects with a prior history of asthma are eligible if they have a current diagnosis of COPD).
* Subjects with alpha1-antitrypsin deficiency as the underlying cause of COPD.
* Subjects with active tuberculosis, lung cancer, and clinically significant: bronchiectasis, sarcoidosis, lung fibrosis, pulmonary hypertension, interstitial lung disease or other active pulmonary diseases.
* Subjects who have undergone lung volume reduction surgery within the 12 months prior to Screening.
* Immune suppression (e.g. advanced human immunodeficiency virus [HIV] with high viral load and low cluster of differentiation 4 [CD4] count, lupus on immunosuppressant's) that in the opinion of the investigator would increase risk of pneumonia or other risk factors for pneumonia (e.g. neurological disorders affecting control of the upper airway, such as Parkinson's Disease, Myasthenia Gravis). Subjects at potentially high risk for pneumonia (e.g. very low body mass index [BMI], severely malnourished, or very low FEV1) will only be included at the discretion of the Investigator.
* Pneumonia and/or moderate or severe COPD exacerbation that has not resolved at least 14 days prior to Screening and at least 30 days following the last dose of oral/systemic corticosteroids (if applicable).
* Respiratory tract infection that has not resolved at least 7 days prior to Screening.
* Chest x-ray (posteroanterior and lateral) reveals evidence of pneumonia or a clinically significant abnormality not believed to be due to the presence of COPD, or another condition that would hinder the ability to detect an infiltrate on chest x-ray (e.g. significant cardiomegaly, pleural effusion or scarring). All subjects will have a chest x-ray at Screening Visit 1 (or historical radiograph or computerized tomography [CT] scan obtained within 3 months prior to screening). For sites in Germany: If a chest x-ray (or CT scan) within 3 months prior to Screening (Visit 1) is not available, approval to conduct a diagnostic chest x-ray will need to be obtained from the Federal Office for Radiation Protection (BfS).
* Subjects with historical or current evidence of clinically significant cardiovascular, neurological, psychiatric, renal, hepatic, immunological, gastrointestinal, urogenital, nervous system, musculoskeletal, skin, sensory, endocrine (including uncontrolled diabetes or thyroid disease) or hematological abnormalities that are uncontrolled. Significant is defined as any disease that, in the opinion of the Investigator, would put the safety of the subject at risk through participation, or which would affect the efficacy or safety analysis if the disease/condition exacerbated during the study.
* Alanine Transaminase (ALT) >2x Upper Limit of Normal (ULN); and bilirubin >1.5x ULN (isolated bilirubin >1.5xULN is acceptable if bilirubin is fractionated and direct bilirubin <35 percent). Current active liver or biliary disease (with the exception of Gilbert's syndrome or asymptomatic gallstones or otherwise stable chronic liver disease per investigator assessment). Chronic stable hepatitis B and C (e.g., presence of hepatitis B surface antigen [HBsAg] or positive hepatitis C antibody test result at screening or within 3 months prior to first dose of study treatment) are acceptable if subject otherwise meets entry criteria.
* Subjects with any of the following at Screening (Visit 1): myocardial infarction or unstable angina in the last 6 months; unstable or life threatening cardiac arrhythmia requiring intervention in the last 3 months; New York Heart Association (NYHA) Class IV Heart failure.
* Abnormal and clinically significant 12-lead electrocardiogram (ECG) finding at Visit 1. The Investigator will determine the clinical significance of each abnormal ECG finding in relation to the Subject's medical history and exclude subjects who would be at undue risk by participating in the trial. An abnormal and clinically significant finding that would preclude a subject from entering the trial is defined as a 12-lead ECG tracing that is interpreted at, but not limited to, any of the following: atrial fibrillation (AF) with rapid ventricular rate >120 beats per minute (BPM); sustained and non-sustained ventricular tachycardia (VT); second degree heart block Mobitz type II and third degree heart block (unless pacemaker or defibrillator had been inserted); QT interval corrected for heart rate (QTc) >=500 millisecond (msec) in subjects with QRS <120 msec and QTc >=530 msec in subjects with QRS >=120 msec.
* A history of allergy or hypersensitivity to any corticosteroid, anticholinergic/muscarinic receptor antagonist, beta2-agonist, lactose/milk protein or magnesium stearate or a medical condition such as narrow-angle glaucoma, prostatic hypertrophy or bladder neck obstruction that, in the opinion of the Investigator, contraindicates study participation.
* Subjects with carcinoma that has not been in complete remission for at least 3 years. Subjects who have had carcinoma in situ of the cervix, squamous cell carcinoma and basal cell carcinoma of the skin would not be excluded based on the 3 year waiting period if the subject has been considered cured by treatment.
* Use of long-term oxygen therapy (LTOT) described as resting oxygen therapy >3 Liters per minute (L/minute) (Oxygen use <=3 L/minute flow is not exclusionary.)
* Subjects who are medically unable to withhold their albuterol/salbutamol for the 4-hour period required prior to spirometry testing at each study visit.
* Subjects who have participated in the acute phase of a Pulmonary Rehabilitation Programme within 4 weeks prior to screening or subjects who plan to enter the acute phase of a Pulmonary Rehabilitation Programme during the study. Subjects who are in the maintenance phase of a Pulmonary Rehabilitation Programme are not excluded.
* Subjects with a known or suspected history of alcohol or drug abuse within the last 2 years.
* Subjects at risk of non-compliance, or unable to comply with the study procedures. Any infirmity, disability, or geographic location that would limit compliance for scheduled visits.
* Subjects with a history of psychiatric disease, intellectual deficiency, poor motivation or other conditions that will limit the validity of informed consent to participate in the study.
* Study Investigators, sub-Investigators, study coordinators, employees of a participating Investigator or study site, or immediate family members of the aforementioned that is involved with this study.
* In the opinion of the Investigator, any subject who is unable to read and/or would not be able to complete study related materials.
* Subjects taking following drug therapies will be excluded; subjects taking inhaled short-acting anticholinergics alone or along with short-acting beta agonist combination within 6 hours prior to screening; subjects taking inhaled short-acting beta2 agonists within >=4 hours prior to screening; subjects taking ICS, ICS/inhaled LABA combinations (e.g., FF/salmeterol, mometasone furoate/formoterol fumarate, budesonide/formoterol fumarate; FF/VI), Phosphodiesterase 4 (PDE4) inhibitors (roflumilast), LABA (e.g., indacaterol, olodaterol), LAMA (e.g., LAMA/LABA combinations UMEC, aclidinium, glycopyrronium), LAMA/LABA combinations, theophyllines, sodium cromoglycate and nedocromil sodium, anti-leukotrienes as maintenance treatment within 3 months prior to Visit 1 will be excluded. Maintenance treatment is defined as use for >=14 consecutive days (at any time in the 3 months prior to Visit 1). Subjects taking long term antibiotic therapy. (Antibiotics are allowed for the short term treatment (<=14 days) of an exacerbation or for short term treatment (<=14 days) of other acute infections during the study); subjects taking systemic, oral, parenteral corticosteroids 30 days prior to screening; (During the study oral/systemic corticosteroids may be used for <=14 days to treat COPD exacerbations/pneumonia) will be excluded. Intra-articular injections are allowed; subjects taking any other investigational drug within 30 days or 5 half-lives whichever is longer prior to screening will be excluded.

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 800 (Actual)
Dates: Start 2018-03-29 (Actual); Primary Completion 2019-07-17 (Actual); Study Completion 2019-07-17 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (62):
- United States (32):
  - GSK Investigational Site, Andalusia, Alabama
  - GSK Investigational Site, Huntington Beach, California
  - GSK Investigational Site, Sacramento, California
  - GSK Investigational Site, Simi Valley, California
  - GSK Investigational Site, Colorado Springs, Colorado
  - GSK Investigational Site, Daytona Beach, Florida
  - GSK Investigational Site, Kissimmee, Florida
  - GSK Investigational Site, Miami, Florida
  - GSK Investigational Site, Miami Lakes, Florida
  - GSK Investigational Site, Orlando, Florida
  - GSK Investigational Site, Ormond Beach, Florida
  - GSK Investigational Site, Panama City, Florida
  - GSK Investigational Site, Nampa, Idaho
  - GSK Investigational Site, Oxon Hill, Maryland
  - GSK Investigational Site, Edina, Minnesota
  - GSK Investigational Site, Minneapolis, Minnesota
  - GSK Investigational Site, Bronxville, New York
  - GSK Investigational Site, Fayetteville, New York
  - GSK Investigational Site, Gastonia, North Carolina
  - GSK Investigational Site, Cincinnati, Ohio
  - GSK Investigational Site, Dublin, Ohio
  - GSK Investigational Site, DuBois, Pennsylvania
  - GSK Investigational Site, Anderson, South Carolina
  - GSK Investigational Site, Gaffney, South Carolina
  - GSK Investigational Site, Greer, South Carolina
  - GSK Investigational Site, Little River, South Carolina
  - GSK Investigational Site, Pelzer, South Carolina
  - GSK Investigational Site, Seneca, South Carolina
  - GSK Investigational Site, Spartanburg, South Carolina
  - GSK Investigational Site, Corsicana, Texas
  - GSK Investigational Site, Huntsville, Texas
  - GSK Investigational Site, Salt Lake City, Utah
- Poland (22):
  - GSK Investigational Site, Bialystok
  - GSK Investigational Site, Bielsko-Biala
  - GSK Investigational Site, Bydgoszcz
  - GSK Investigational Site, Chojnice
  - GSK Investigational Site, Grudziądz
  - GSK Investigational Site, Kielce
  - GSK Investigational Site, Krakow
  - GSK Investigational Site, Lublin
  - GSK Investigational Site, Nowa Sól
  - GSK Investigational Site, Ostrowiec Świętokrzyski
  - GSK Investigational Site, Ostróda
  - GSK Investigational Site, Piaseczno
  - GSK Investigational Site, Proszowice
  - GSK Investigational Site, Siedlce
  - GSK Investigational Site, Skierniewice
  - GSK Investigational Site, Sopot
  - GSK Investigational Site, Swidnica
  - GSK Investigational Site, Szczecin
  - GSK Investigational Site, Torun
  - GSK Investigational Site, Warsaw
  - GSK Investigational Site, Zamość
  - GSK Investigational Site, Zawadzkie
- Russia (8):
  - GSK Investigational Site, Ivanovo
  - GSK Investigational Site, Moscow
  - GSK Investigational Site, Novosibirsk
  - GSK Investigational Site, Saint Petersburg
  - GSK Investigational Site, Saratov
  - GSK Investigational Site, Ulyanovsk
  - GSK Investigational Site, Voronezh
  - GSK Investigational Site, Yekaterinburg

IPD SHARING:
Plan to Share IPD: Yes
IPD for this study is available via the Clinical Study Data Request site
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: IPD is available via the Clinical Study Data Request site (copy the URL below to your browser)
Access Criteria: Access is provided after a research proposal is submitted and has received approval from the Independent Review Panel and after a Data Sharing Agreement is in place. Access is provided for an initial period of 12 months but an extension can be granted, when justified, for up to another 12 months.
URL: https://www.clinicalstudydatarequest.com/Posting.aspx?ID=20851

REFERENCES:
- [Background] Bansal S, Anderson M, Anzueto A, Brown N, Compton C, Corbridge TC, Erb D, Harvey C, Kaisermann MC, Kaye M, Lipson DA, Martin N, Zhu CQ, Papi A. Single-inhaler fluticasone furoate/umeclidinium/vilanterol (FF/UMEC/VI) triple therapy versus tiotropium monotherapy in patients with COPD. NPJ Prim Care Respir Med. 2021 May 25;31(1):29. doi: 10.1038/s41533-021-00241-z. PMID 34035312

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This was a randomized, multicenter, parallel group study where participants with chronic obstructive pulmonary disease (COPD) were randomized to receive either fluticasone furoate/umeclidinium/vilanterol or tiotropium in a 1:1 ratio. The study was conducted across 68 centers in 3 countries.
Pre-assignment Details: A total of 1049 participants were screened, of which 179 failed screening. Total of 870 participants entered in run-in period, of which 70 were run-in failures. Total of 800 participants were enrolled and randomized.
Groups:
- Fluticasone Furoate/Umeclidinium/Vilanterol 100/62.5/25 mcg: Participants received fluticasone furoate/umeclidinium/vilanterol (FF/UMEC/VI) 100/62.5/25 microgram (mcg) via the ELLIPTA (once daily in the morning) plus placebo to match tiotropium (TIO) via HandiHaler (once daily in the morning) for 84 days. Participants received albuterol/salbutamol as rescue medication via metered dose inhaler (MDI) during conduct of the study, if required.
- Tiotropium 18 mcg: Participants received tiotropium 18 mcg via HandiHaler (once daily in the morning) plus placebo to match fluticasone furoate/umeclidinium/vilanterol via the ELLIPTA (once daily in the morning) for 84 days. Participants received albuterol/salbutamol as rescue medication via MDI during conduct of the study, if required.
Period: Overall Study
Arm/Group | Fluticasone Furoate/Umeclidinium/Vilanterol 100/62.5/25 mcg | Tiotropium 18 mcg
Started | 400 | 400
Received Study Treatment | 400 | 399 (One randomized participant withdrew consent and never received study treatment.)
Completed | 383 | 387
Not Completed | 17 | 13
Not completed — Adverse Event | 6 | 3
Not completed — Lost to Follow-up | 2 | 1
Not completed — Physician Decision | 3 | 2
Not completed — Withdrawal by Subject | 5 | 7
Not completed — Investigator site closed | 1 | 0

BASELINE CHARACTERISTICS:
Population: Baseline characteristics were presented for all randomized participants including one randomized participant who withdrew consent and never received study treatment in "Tiotropium 18 mcg" arm.
Groups:
- Total: Total of all reporting groups
Arm/Group | Fluticasone Furoate/Umeclidinium/Vilanterol 100/62.5/25 mcg | Tiotropium 18 mcg | Total
Number analyzed (Participants) | 400 | 400 | 800
Age, Continuous [Mean (Standard Deviation); unit: Years] | 66.2 (8.08) | 66.1 (7.78) | 66.2 (7.93)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 126 | 131 | 257
  Male | 274 | 269 | 543
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  African American/African Heritage | 10 | 12 | 22
  White - White/Caucasian/European Heritage | 390 | 388 | 778

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Trough Forced Expiratory Volume in 1 Second (FEV1) on Day 85
Description: FEV1 is a measure of lung function and is defined as the maximal amount of air that can be forcefully exhaled in one second. Trough FEV1 on Day 85 was defined as the mean of the two planned spirometry FEV1 measurements. Change from Baseline in trough FEV1 on Day 85 was calculated by subtracting Baseline FEV1 value from the trough FEV1 value on Day 85. Baseline FEV1 was defined as the mean of the two assessments made at 30 and 5 minutes pre-dose on Day 1.
Time Frame: Baseline (Day 1 [Pre-dose at 30 minutes and 5 minutes]) and Day 85
Population: Intent-To-Treat (ITT) Population comprised of all randomized participants, excluding those who were randomized in error. Only those participants with data available at the specified time point were analyzed.
Measure: Least Squares Mean (Standard Error); unit: Liters
Arm/Group | Fluticasone Furoate/Umeclidinium/Vilanterol 100/62.5/25 mcg | Tiotropium 18 mcg
Number analyzed (Participants) | 362 | 375
Liters | 0.115 (0.0119) | 0.020 (0.0117)
Statistical Analysis 1: Comparison: Fluticasone Furoate/Umeclidinium/Vilanterol 100/62.5/25 mcg vs Tiotropium 18 mcg; Test type: Superiority; p < 0.001, Mixed model repeated measures (MMRM) — The MMRM model included Baseline FEV1, visit, geographical region, and treatment as covariates and visit-by-Baseline FEV1 and visit-by-treatment interaction terms; Mean Difference (Net) = 0.095, 95% CI 2-sided [0.062 to 0.128], Standard Error of Mean 0.0167

2. Secondary Outcome: Change From Baseline in Trough FEV1 on Day 28
Description: FEV1 is a measure of lung function and is defined as the maximal amount of air that can be forcefully exhaled in one second. Trough FEV1 on Day 28 was defined as the average of the two pre-dose FEV1 measurements recorded before the morning dose of randomized study medication on Day 28. Change from Baseline in trough FEV1 on Day 28 was calculated by subtracting Baseline FEV1 value from the trough FEV1 value on Day 28. Baseline FEV1 was defined as the mean of the two assessments made at 30 and 5 minutes pre-dose on Day 1.
Time Frame: Baseline (Day 1 [Pre-dose at 30 minutes and 5 minutes]) and Day 28
Population: ITT Population. Only those participants with data available at the specified time point were analyzed.
Measure: Least Squares Mean (Standard Error); unit: Liters
Arm/Group | Fluticasone Furoate/Umeclidinium/Vilanterol 100/62.5/25 mcg | Tiotropium 18 mcg
Number analyzed (Participants) | 385 | 390
Liters | 0.115 (0.0102) | -0.007 (0.0101)
Statistical Analysis 1: Comparison: Fluticasone Furoate/Umeclidinium/Vilanterol 100/62.5/25 mcg vs Tiotropium 18 mcg; Test type: Superiority; p < 0.001, Mixed model repeated measures (MMRM) — [p-value comment as in outcome 1, analysis 1]; Mean Difference (Net) = 0.122, 95% CI 2-sided [0.094 to 0.150], Standard Error of Mean 0.0144

3. Secondary Outcome: Change From Baseline in Trough FEV1 on Day 84
Description: FEV1 is a measure of lung function and is defined as the maximal amount of air that can be forcefully exhaled in one second. Trough FEV1 on Day 84 was defined as the average of the two pre-dose FEV1 measurements recorded before the morning dose of randomized study medication on Day 84. Change from Baseline in trough FEV1 on Day 84 was calculated by subtracting Baseline FEV1 value from the trough FEV1 value on Day 84. Baseline FEV1 was defined as the mean of the two assessments made at 30 and 5 minutes pre-dose on Day 1.
Time Frame: Baseline (Day 1 [Pre-dose at 30 minutes and 5 minutes]) and Day 84
Population: ITT Population. Only those participants with data available at the specified time point were analyzed.
Measure: Least Squares Mean (Standard Error); unit: Liters
Arm/Group | Fluticasone Furoate/Umeclidinium/Vilanterol 100/62.5/25 mcg | Tiotropium 18 mcg
Number analyzed (Participants) | 376 | 386
Liters | 0.105 (0.0113) | 0.018 (0.0111)
Statistical Analysis 1: Comparison: Fluticasone Furoate/Umeclidinium/Vilanterol 100/62.5/25 mcg vs Tiotropium 18 mcg; Test type: Superiority; p < 0.001, Mixed model repeated measures (MMRM) — [p-value comment as in outcome 1, analysis 1]; Mean Difference (Net) = 0.087, 95% CI 2-sided [0.056 to 0.118], Standard Error of Mean 0.0159

4. Secondary Outcome: Number of Participants With Non-serious Adverse Events (Non-SAEs) and Serious Adverse Events (SAEs)
Description: An AE is any untoward medical occurrence in a clinical study participant, temporally associated with the use of a study treatment, whether or not considered related to the study treatment. Any untoward event resulting in death, life threatening, requires hospitalization or prolongation of existing hospitalization, results in disability/incapacity, congenital anomaly/birth defect or any other important medical event according to medical or scientific judgement was categorized as SAE.
Time Frame: Up to Day 95
Population: ITT Population. Non-SAEs and SAEs were presented for all randomized participants excluding one participant in ITT population who was randomized correctly to "Tiotropium 18 mcg" arm but did not take any randomized study treatment due to withdrawal of consent.
Measure: Count of Participants; unit: Participants
Arm/Group | Fluticasone Furoate/Umeclidinium/Vilanterol 100/62.5/25 mcg | Tiotropium 18 mcg
Number analyzed (Participants) | 400 | 399
Participants
  Non-SAEs | 31 | 29
  SAEs | 13 | 11

5. Secondary Outcome: Change From Baseline in Systolic Blood Pressure (SBP) and Diastolic Blood Pressure (DBP)
Description: SBP and DBP were assessed in the sitting position after approximately 5 minutes rest. Change from Baseline was calculated by subtracting Baseline value from the post-dose visit value. Baseline was defined as the latest pre-first-dose assessment with a non-missing value, including those from unscheduled visits.
Time Frame: Baseline (Day 1, Pre-dose) and Day 84
Population: ITT Population. Only those participants with data available at the specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: Millimeters of mercury
Arm/Group | Fluticasone Furoate/Umeclidinium/Vilanterol 100/62.5/25 mcg | Tiotropium 18 mcg
Number analyzed (Participants) | 387 | 392
Millimeters of mercury
  SBP | -0.3 (12.53) | -0.1 (11.02)
  DBP | -0.3 (8.17) | -0.7 (7.88)

6. Secondary Outcome: Change From Baseline in Pulse Rate
Description: Pulse rate was assessed in the sitting position after approximately 5 minutes rest. Change from Baseline was calculated by subtracting Baseline value from the post-dose visit value. Baseline was defined as the latest pre-first-dose assessment with a non-missing value, including those from unscheduled visits.
Time Frame: Baseline (Day 1, Pre-dose) and Day 84
Population: ITT Population. Only those participants with data available at the specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: Beats per minute
Arm/Group | Fluticasone Furoate/Umeclidinium/Vilanterol 100/62.5/25 mcg | Tiotropium 18 mcg
Number analyzed (Participants) | 387 | 392
Beats per minute | 0.2 (8.55) | 0.8 (8.51)

ADVERSE EVENTS:
Time Frame: Non-SAEs and SAEs were reported from start of study treatment and up to 95 days
Description: Non-SAEs and SAEs were presented for all randomized participants excluding one randomized participant who withdrew consent and never received study treatment in "Tiotropium 18 mcg" arm. Adverse events were presented treatment-wise.
Arm/Group | Fluticasone Furoate/Umeclidinium/Vilanterol 100/62.5/25 mcg | Tiotropium 18 mcg
All-Cause Mortality (participants affected / at risk) | 2/400 | 1/399
Serious Adverse Events (participants affected / at risk) | 13/400 | 11/399
Other Adverse Events (participants affected / at risk) | 31/400 | 29/399
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Fluticasone Furoate/Umeclidinium/Vilanterol 100/62.5/25 mcg (N=400) | Tiotropium 18 mcg (N=399)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 1 (1)
Cardiac arrest (Cardiac disorders) | 1 (1) | 0 (0)
Cardiac failure (Cardiac disorders) | 1 (1) | 0 (0)
Pancreatitis acute (Gastrointestinal disorders) | 1 (1) | 1 (1)
Small intestinal obstruction (Gastrointestinal disorders) | 1 (1) | 1 (1)
Cholecystitis acute (Hepatobiliary disorders) | 0 (0) | 1 (1)
Cholelithiasis (Hepatobiliary disorders) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 1 (1) | 3 (3)
Postoperative wound infection (Infections and infestations) | 1 (1) | 0 (0)
Diabetes mellitus inadequate control (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Rheumatoid arthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Haemorrhagic stroke (Nervous system disorders) | 0 (0) | 1 (1)
Ischaemic stroke (Nervous system disorders) | 0 (0) | 1 (1)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 5 (6) | 3 (3)
Angioedema (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Fluticasone Furoate/Umeclidinium/Vilanterol 100/62.5/25 mcg (N=400) | Tiotropium 18 mcg (N=399)
Headache (Nervous system disorders) | 18 (30) | 22 (69)
Nasopharyngitis (Infections and infestations) | 16 (17) | 8 (8)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.

DOCUMENTS (2):
  • Study Protocol (2018-07-17): https://cdn.clinicaltrials.gov/large-docs/81/NCT03474081/Prot_000.pdf
  • Statistical Analysis Plan (2019-07-30): https://cdn.clinicaltrials.gov/large-docs/81/NCT03474081/SAP_001.pdf